CLINICAL TRIAL: NCT06650605
Title: Citadel-123: a Phase I Clinical Trial to Assess the Activity of I-123 Poly Adenosine Diphosphate Ribose Polymerase I Inhibitor (123I-ATT001) Directly Administered in Subjects with Relapsed Glioblastoma.
Brief Title: Phase 1 Open-label Study of 123I-ATT001 in Subjects with Relapsed Glioblastoma
Acronym: CITADEL-123
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Theragnostics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIL101; 1006521 (Other: IRAS)
Record Dates: First submitted 2024-07-16; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Glioma Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Part 1 Dose Escalation & Dose Expansion (Experimental): Dose Escalation:
  123I-ATT001 Dose Level 1 123I-ATT001 Dose Level 2 123I-ATT001 Dose Level 3
  Dose Expansion:
  123I-ATT001 Recommended Dose from Dose Escalation
  Interventions: Drug: 123I-ATT001

INTERVENTIONS:
Drug: 123I-ATT001 — 123I-ATT001

SUMMARY:
Phase I open-label trial of 123I-ATT001 monotherapy and in combination with treatment therapies in subjects with relapsed glioblastoma.

DETAILED DESCRIPTION:
The main goals of this study are to understand if 123I-ATT001 is safe and tolerable to treat participants with relapsed glioblastoma and to determine the maximum tolerated dose that can be given to participants without any unacceptable side effects.

The study consists of two parts:

- Part 1 is a dose escalation study where three doses of 123I-ATT001 will be tested, starting with the lowest dose. When a recommended dose (RD) has been declared, a monotherapy expansion cohort will be open at that dose level.

In Part 1 participants will receive a 123I-ATT001 dose, once per week, for four weeks (+ two optional extra cycles).

* Part 2 is a dose expansion study where one dose of 123I-AT001 will be tested in combination with other therapies. Part 2 will begin after the Part 1 has completed and a recommended part 2 dose has been chosen.

The specific details and combination therapies for Part 2 of the study will be added via a protocol amendment at a later date.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent
2. Men and women over 18 years of age.
3. Histologically confirmed recurrent glioblastoma (grade IV) as per WHO criteria 2021 (IDH- wild type only) where the subjects have an Ommaya reservoir in an intralesional cavity of at least 5 mL volume.
4. Documented recurrent disease (radiological, based on RANO v.1.0) within 3 months prior to first study drug administration with no suitable standard of care options available.
5. Eastern Cooperative Oncology Group Performance status of 0 or 1.
6. Adequate organ function
7. Women of childbearing potential must use two forms of reliable contraception before starting 123I-ATT001 treatment, during therapy and for 6 months after receiving the last dose of 123I-ATT001. All male subjects must agree to not donate sperm during the study and for 6 months after the last dose of study drug.
8. Be able to understand and comply with the requirements of the study, as judged by the Investigator.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Diagnosis of immunodeficiency or receiving systemic steroid therapy of up to 4 mg/ day dexamethasone or equivalent or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
3. Prior anticancer treatments within the following time periods:

   1. Chemotherapy within 4 weeks of enrolment or 5 half-lives, whichever is shorter.
   2. Targeted small molecule therapy within 4 weeks of enrolment or 5 half-lives, whichever is shorter.
   3. Immunotherapy (including monoclonal antibody therapy) or radiation therapy within 4 weeks prior to study day 1.
4. Unresolved NCI-CTCAE grade 2 or higher toxicity (except stable neurological toxicities/deficits related to disease process, alopecia).
5. Patients with a known allergy to Olaparib or Iodine.
6. Known additional malignancy that is progressing or requires active treatment excepting basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
7. Any condition that precludes the proper performance of SPECT and/or MRI scan
8. Any clinically significant abnormalities in resting ECG at the time of screening including prolonged QTcF (>450 ms for males; >470 ms for females) and cardiac arrhythmias, as judged by the Investigator or designee.
9. Unstable systemic disease (including but not limited to active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
10. Psychiatric, substance misuse or functional disorders that prevent subjects from providing informed consent, following protocol instructions or cooperating with the requirements of the study.
11. Active infection requiring systemic therapy.
12. Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the pre-screening or screening visit through 3 months after the last dose of study treatment.
13. Subject that has a condition or is in a situation, which in the Investigators opinion may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.
14. History of non- infectious pneumonitis within the last 3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Dose Escalation: Frequency and severity of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | Screening to end of treatment visit (28 days after last dose of 123I-ATT001)
  To assess safety and tolerability of 123I-ATT001
Part 1- Dose Escalation: Incidence of Dose Limiting Toxicity (DLT) | Day 1 to Day 14 of 123I-ATT001 administration
  Evaluated by monitoring of Adverse Events.

SECONDARY OUTCOMES:
Part 1 - Dose Escalation: biodistribution and pharmacokinetics of 123I-ATT001 in blood | Collected 1 hour, 4 hours and 24 hours post each dose and optionally at 48 hours post first dose.
  Blood samples will be collected from the first 6 patients in Part 1.
Part 1- Dose Escalation: biodistribution and pharmacokinetics of 123I-ATT001 in urine. | Collected 24 hours post first dose
  Urine samples will be collected from the first 6 patients in Part 1.
Part 1 - Dose Escalation: radiation dosimetry of 123I-ATT001 (exposure of each organ to radiation) | 1 and 4 and 24 hours post first dose and 4 hours post fourth dose.
  SPECT/CT and or whole body planar imaging
Part 1- Dose Escalation: preliminary assessment of the antitumour activity of 123I-ATT001 | Screening, Day 14 post each dose, 28 days after last dose, then a further 3 times every 8 weeks at follow up.
  Efficacy will be assessed according to the RANO response criteria using MRI Scans
Part 1 - Dose Escalation: effect of 123I-ATT001 on neurological function | Screening, the day of the 1st, 3rd and 5th (if given) dose, may also be performed within 48 hours prior to dose administration. It will also be performed on the End of Treatment visit which takes place 28 days post last dose.
  Neurological function will be assessed by the principal investigator according to NANO criteria.
Part 1 - Dose Escalation: effect of 123I-ATT001 on neurological function | Screening, the day of the 1st, 3rd and 5th (if given) dose, may also be performed within 48 hours prior to dose administration. It will also be performed on the End of Treatment visit which takes place 28 days post last dose.
  Patients will complete the MDASI-BT questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mulholland, Principal Investigator — University College London Hospital
Locations (2):
- United Kingdom (2):
  - University College London Hosptial, London
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No
no current plans to share any data with other researcheers

REFERENCES:
- See also: Related Info — https://ariceum-therapeutics.com/pipeline/rparpi/